CLINICAL TRIAL: NCT00347191
Title: Phase 4 Study Evaluating the Relationship Between Intraocular Pressure and Central Corneal Thickness Using Various Instruments in Ocular Hypertension, Normal-tension Glaucoma, Primary Open Angle Glaucoma, Keratoconus and Normal Eyes.
Brief Title: Relationship Between Central Corneal Thickness and Intraocular Pressure Measures Instruments.
Status: Completed | Type: Observational
Sponsor: Aston University (Other)
Other Study IDs: 2006IOP
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Glaucoma; Glaucoma, Open Angle; Ocular Hypertension; Keratoconus
Keywords: Corneal thickness; Intraocular pressure; Instrumentation; Glaucoma; Keratoconus
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle; Ocular Hypertension; Keratoconus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the relationship between intraocular pressure and central corneal thickness using various instruments in ocular hypertension, normal-tension glaucoma, primary open angle glaucoma, keratoconus and normal eyes.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the relationship between intraocular pressure and ultrasound pachymetry measured central corneal thickness using Goldman tonometry and PASCAL instruments.

Patient groups examined include:

ocular hypertensives normal-tension glaucoma primary open angle glaucoma keratoconus control normal eyes

ELIGIBILITY:
Inclusion Criteria:

Adults over the age of 18 years Clinical diagnosis of glaucoma, open angle; ocular hypertension; glaucoma (low-tension); keratoconus and other healthy volunteers.

Exclusion Criteria:

Children under the age of 18 years Adults with learning disabilities Adults who are unconscious or severely ill Adults who have known terminal illness Adults in emergency situations Adults with dementia Prisoners Young offenders Those who could be considered to have a dependant relationship with the investigator (i.e. those in care homes or medical students) Other vulnerable groups

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinical diagnosis of glaucoma, open angle; ocular hypertension; glaucoma (low-tension); keratoconus and other healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 1000
Dates: Start 2006-01; Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Shah, MD FRCOphth, Principal Investigator — Birmingham and Midland Eye Centre
Locations (1):
- Solihull Hospital, Birmingham, West Midlands, United Kingdom